CLINICAL TRIAL: NCT03928210
Title: Effect of Digoxin on Clusters of Circulating Tumor Cells (CTCs) in Breast Cancer Patients
Brief Title: Digoxin Induced Dissolution of CTC Clusters
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ETH Zurich - The Aceto Lab (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00673; sp19Kurzeder
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Circulating Tumor Cells (CTCs)
Keywords: cluster of circulating tumor cells (CTCs); cardiac glycosides; digoxin
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Digoxin

STUDY DESIGN:
Intervention Model Description: Patients with at least one CTC cluster (if homotypic ≥ 2 CTCs, if heterotypic ≥ 1 CTC and ≥ 1 white blood cell (WBC)) at screening entered the treatment phase. During treatment phase, patients received a daily maintenance dose of digoxin for a total of seven days, with a digoxin target level of ≥ 0.7 ng/ml in serum during treatment. Blood draws for capture and enumeration of CTCs and CTC clusters were obtained on day 0 (pre- and 2 hours post digoxin), day 3 and day 7. Regular study visits included clinical and laboratory assessments such as vital signs, electrocardiogram (ECG), serious adverse events (SAE), and digoxin serum levels on day 0 and 7.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digoxin (Experimental): Digoxin 0.125 mg or 0.25 mg administered once daily for 7 days or until symptoms of toxicity Generic e.g. DIGOXIN Juvisé or Lenoxin Mite
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin — Patients will receive a daily maintenance dose of digoxin. The daily dose of digoxin will be calculated according to the renal function and the target serum digoxin concentration and applied in an adjusted regimen based on the availability of 0.125 mg and 0.25 mg pills in the morning (before 10 am). Blood samples for analyses of mean CTC cluster size will be drawn at screening, on day 0 (2 hrs after first oral intake), on day 3 and on day 7. Depending on the digoxin serum level maintenance therapy with digoxin will be continued up to 3 weeks if the digoxin serum level on day 7 or day 14 is below 0.70 ng/ml. For the third week of maintenance therapy individual dose adjustments will be carried out as needed.
  Other Names: Lenoxin Mite; DIGOXIN Juvisé

SUMMARY:
This single arm therapeutic exploratory study of digoxin in patients with advanced or metastatic breast cancer investigates whether cardiac glycosides are able to disrupt CTC clusters in breast cancer patients.

DETAILED DESCRIPTION:
Circulating tumor cells (CTCs) are considered to be precursors of metastasis in various cancer types and are found in the blood of cancer patients as single CTCs and CTC clusters, with the latter featuring a higher ability to seed metastasis.

CTC cluster share several properties that commonly feature stem cell biology which drive metastases formation. Preclinical data shows that CTC clusters can be disaggregated into single cells by the treatment with cardiac glycosides such as digoxin. This single arm therapeutic exploratory study of digoxin in patients with advanced or metastatic breast cancer investigates whether cardiac glycosides are able to disrupt CTC clusters in breast cancer patients.

Patients with advanced or metastatic breast cancer in whom CTC clusters could be identified will receive an individualized daily maintenance dose of digoxin adapted to their kidney function. Blood samples for analyses of digoxin serum level and mean CTC cluster size will be drawn at specified time points.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Diagnosis of adenocarcinoma of the breast with evidence of locoregionally recurrent or metastatic disease not amenable to resection, radiation therapy or systemic therapy with curative intent
* Adequate organ and marrow function

Exclusion Criteria:

* Patients on treatment with digoxin or digitoxin
* Patients with atrial fibrillation or atrial flutter
* Ventricular Fibrillation or ventricular tachycardia,
* Atrioventricular heart block 2nd or 3rd degree, sick sinus syndrome or sinus bradycardia,
* Wolff-Parkinson-White Syndrome
* Hypokalemia, hypercalcemia, hypomagnesemia, hypoxia,
* Hypertrophic cardiomyopathy, aortic aneurysm
* Simultaneous intravenous application of calcium salts
* Known hypersensitivity to Digoxin, other cardiac glycosides or included compounds
* Known drug interactions of ongoing cancer therapy with digoxin
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in mean CTC cluster size (in ng/ml) | Blood samples drawn at Screening, on day 0 (2 hours after first oral intake of digoxin), on day 3, on day 7, on day 10, on day 14, on day 17 and on day 21 after first oral intake of digoxin
  mean CTC cluster size (in patients with a digoxin serum level above 0.7 ng/ml) after treatment will be compared to mean CTC-cluster size before treatment

SECONDARY OUTCOMES:
Change in mean CTC cluster number | Blood samples drawn at Screening, on day 0 (2 hours after first oral intake of digoxin), on day 3, on day 7, on day 10, on day 14, on day 17 and on day 21 after first oral intake of digoxin
  number of CTC-clusters before and after treatment will be compared
Average time to dissolution of CTC Clusters (in days) | Blood samples drawn at Screening, on day 0 (2 hours after first oral intake of digoxin), on day 3, on day 7, on day 10, on day 14, on day 17 and on day 21 after first oral intake of digoxin
  average time to dissolution of CTC clusters

CONTACTS AND LOCATIONS:
Overall Officials: Christian Kurzeder, PD Dr. med, Principal Investigator — Breast Cancer Center, University Hospital Basel
Locations (3):
- Switzerland (3):
  - Kantonspital Baselland (KSBL), Liestal, Basel-Landschaft
  - Breast Cancer Center, University Hospital Basel, Basel
  - University Hospital Zurich (USZ), Zurich

REFERENCES:
- [Derived] Kurzeder C, Nguyen-Strauli BD, Krol I, Ring A, Castro-Giner F, Nuesch M, Asawa S, Zhang YW, Budinjas S, Gvozdenovic A, Vogel M, Kohler A, Grasic Kuhar C, Schwab FD, Heinzelmann-Schwarz V, Weber WP, Rochlitz C, Vorburger D, Frauchiger-Heuer H, Witzel I, Wicki A, Kuster GM, Vetter M, Aceto N. Digoxin for reduction of circulating tumor cell cluster size in metastatic breast cancer: a proof-of-concept trial. Nat Med. 2025 Apr;31(4):1120-1124. doi: 10.1038/s41591-024-03486-6. Epub 2025 Jan 24. PMID 39856336